CLINICAL TRIAL: NCT06478316
Title: Pain Control With Intracervical Block, During Laminaria Insertion for Late Abortions, a Double Blind Randomized Control Trial
Brief Title: Intracervical Block During Laminaria Insertion
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ASF-0020-24
Record Dates: First submitted 2024-06-16; First posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Late Abortion; Dilation and Evacuation
MeSH Terms: conditions — Dilatation, Pathologic

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study (Experimental): a 10 ml syringe will be filled with 7 ml of lidocaine and 1 ml of bicarbonate (total 70 mg of lidocaine).
  Interventions: Procedure: Intracervical block
- Control (Sham Comparator): a 10 ml syringe will be filled with 8 ml of 0.9% NaCl saline
  Interventions: Procedure: Intracervical block

INTERVENTIONS:
Procedure: Intracervical block — local injection of lidocain to the cervix

SUMMARY:
Whether intracervical block with lidocaine 1% is superior to sham procedure - intracervical injection of saline 0.9% - in terms of pain control.

DETAILED DESCRIPTION:
* Research Design - Double-blind randomized study
* Study Population - Women who are candidates for late termination of pregnancy by dilation and evacuation and approach for the insertion of laminaria will be recruited for the study.
* The women will be divided into two groups

  * Research Group - Women who will undergo preparation for the insertion of laminaria by anesthesia with lidocaine spray, followed by an intracervical injection of 1% lidocaine.
  * Control Group - Women who will be anesthetized with lidocaine spray + intracervical injection of an inactive substance (0.9% saline).
  * Randomization will be performed using dedicated computer software according to blocks of 2-6 women.
* All women will be offered to take 400 mg of ibuprofen about half an hour before the procedure.

  * In the research group - a 10 ml syringe will be filled with 7 ml of lidocaine and 1 ml of bicarbonate (total 70 mg of lidocaine).
  * In the control group - a 10 ml syringe will be filled with 8 ml of 0.9% NaCl saline.
* Primary anesthesia will be performed using 10% lidocaine spray in up to 5 sprays.
* Injection into the cervix will be performed at 3, 6, 9, 12 o'clock positions, after prior aspiration, with a 23-gauge needle, about 2 ml per point.
* Laminaria type to be inserted - "small" diameter 3 mm, length 6.5 cm (MedGyn: Lombard, IL, USA, and Norscan: Westlake Village, CA, USA).

  * At weeks 18-20, 7-9 laminaria will be inserted.
  * Over 20 weeks - over 10 laminaria will be inserted.
* Number of participants in the study - 70.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary termination of pregnancy approved by a committee or missed abortion
* 18.0 to 22.5 gestational week (The gestational age in the case of a missed abortion is determined by the BPD - Biparietal Diameter, which is the determining measure for the ability to perform D&E.)
* Singleton pregnancy

Exclusion Criteria:

* Multiple pregnancy
* Women undergoing the procedure urgently due to cervical insufficiency, inevitable abortion, premature rupture of membranes, or suspected chorioamnionitis
* Allergy to lidocaine
* Women who do not speak Hebrew or English
* Women who have a guardian for any reason
* Women with a history of cesarean section
* Women with abnormal placental implantation, such as placenta previa or suspected placenta accreta
* Women with a psychiatric illness
* Women with a history of alcoholism or drug abuse
* Women who required a "two-stage" laminaria insertion will not be included in the analysis. In cases where the cervix does not allow the insertion of the required number of laminaria, the process is carried out in two stages: in the first stage, the maximum possible number is inserted, the woman is hospitalized, and after a few hours when some initial dilation of the cervix has occurred, the laminaria are removed and new ones are inserted according to the required number

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Pain level using 0-100 Visual Analog Scale (100=worst pain) | During the procedure
  Patients will be asked to rate their maximal pain level during the procedure of laminaria insertion using 0-100 Visual Analog Scale
Rate of patient reporting severe pain (VAS 75-100) during laminaria insertion | During the procedure
  Patients will be asked to rate their maximal pain level during the procedure of laminaria insertion using 0-100 Visual Analog Scale

SECONDARY OUTCOMES:
The rate of complications | During and immediately after the procedure
  Complications during laminaria insertion: rupture of the membranes, cervical bleeding, false route; complication during dilation and evacuation - failure to complete the dilation and evacuation procedure
Acceptability of the procedure measured as the rate of patients who will state that they found the procedure acceptable | Immediately after the procedure
  Patients will be asked to state whether they find the procedure they undergone acceptable

CONTACTS AND LOCATIONS:
Overall Officials: Matan Mor, MD, Principal Investigator — Assaf-Harofeh Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fox MC, Hayes JL; Society of Family Planning. Cervical preparation for second-trimester surgical abortion prior to 20 weeks of gestation. Contraception. 2007 Dec;76(6):486-95. doi: 10.1016/j.contraception.2007.09.004. Epub 2007 Nov 9. PMID 18061709
- [Result] Grimes DA, Schulz KF, Cates WJ Jr. Prevention of uterine perforation during curettage abortion. JAMA. 1984 Apr 27;251(16):2108-11. PMID 6708260
- [Result] Borgatta L, Roncari D, Sonalkar S, Mark A, Hou MY, Finneseth M, Vragovic O. Mifepristone vs. osmotic dilator insertion for cervical preparation prior to surgical abortion at 14-16 weeks: a randomized trial. Contraception. 2012 Nov;86(5):567-71. doi: 10.1016/j.contraception.2012.05.002. Epub 2012 Jun 6. PMID 22682721
- [Result] Prairie BA, Lauria MR, Kapp N, Mackenzie T, Baker ER, George KE. Mifepristone versus laminaria: a randomized controlled trial of cervical ripening in midtrimester termination. Contraception. 2007 Nov;76(5):383-8. doi: 10.1016/j.contraception.2007.07.008. Epub 2007 Oct 4. PMID 17963864
- [Result] Mercier RJ, Liberty A. Intrauterine lidocaine for pain control during laminaria insertion: a randomized controlled trial. Contraception. 2014 Dec;90(6):594-600. doi: 10.1016/j.contraception.2014.07.008. Epub 2014 Jul 23. PMID 25139724
- [Result] Shaw KA, Lerma K. Update on second-trimester surgical abortion. Curr Opin Obstet Gynecol. 2016 Dec;28(6):510-516. doi: 10.1097/GCO.0000000000000318. PMID 27684047
- [Result] Ramesh S, Roston A, Zimmerman L, Patel A, Lichtenberg ES, Chor J. Misoprostol 1 to 3 h preprocedure vs. overnight osmotic dilators prior to early second-trimester surgical abortion. Contraception. 2015 Sep;92(3):234-40. doi: 10.1016/j.contraception.2015.04.005. Epub 2015 Apr 16. PMID 25891258
- [Result] Lerma K, Blumenthal PD. Current and potential methods for second trimester abortion. Best Pract Res Clin Obstet Gynaecol. 2020 Feb;63:24-36. doi: 10.1016/j.bpobgyn.2019.05.006. Epub 2019 May 25. PMID 31281014
- [Result] Creinin MD, Schimmoeller NR, Matulich MC, Hou MY, Melo J, Chen MJ. Gabapentin for pain management after osmotic dilator insertion and prior to dilation and evacuation: A randomized controlled trial. Contraception. 2020 Mar;101(3):167-173. doi: 10.1016/j.contraception.2019.12.001. Epub 2020 Jan 10. PMID 31927028